CLINICAL TRIAL: NCT04542486
Title: Clinical Efficacy of Soft Tissue Trimmer on Postoperative Pain and Wound Healing When Compared to the Conventional Surgical Excision of Gingival Hyperplasia: A Randomized Clinical Trial
Brief Title: Clinical Efficacy of Soft Tissue Trimmer in Cases of Gingival Hyperplasia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Mohamed Sameh, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PER 3-3-1
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Pain, Postoperative; Wound Heal; Gingival Hyperplasia
MeSH Terms: conditions — Pain, Postoperative; Gingival Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The conventional approach: (Experimental): Gingivoplasties and removal of excess gingival tissues through the conventional scalpel technique using a reverse bevel.
  Interventions: Procedure: Excision of gingival hyperplasia using the conventional scalpel technique
- The intervention approach: (Active Comparator): Gingivoplasties and elimination of excess gingival tissues through the use of "Soft tissue trimmer".
  Interventions: Procedure: Excision of gingival hyperplasia using "Soft tissue trimmer ".

INTERVENTIONS:
Procedure: Excision of gingival hyperplasia using "Soft tissue trimmer ". — Gingivoplasties and removal of excess gingival tissues using Soft tissue trimmer.
  Arms: The intervention approach:
Procedure: Excision of gingival hyperplasia using the conventional scalpel technique — Excision of gingival hyperplasia in gingivoplasties using the conventional technique reverse bevel using 15c blade.
  Arms: The conventional approach:

SUMMARY:
Postoperative pain and wound healing are compared after using conventional scalpel technique in comparison with the intervention which is using Soft tissue Trimmer for cases of gingival hyperplasia.

DETAILED DESCRIPTION:
In the control group:

1. Following the local anaesthetic administration, A reverse bevel gingivectomy will be performed with a #15c scalpel.
2. The borderline of gingiva will be determined via the use of a pointer dental tweezers, and excessive gingival tissue will then be removed with Gracey curettes
3. No periodontal packs to be applied to ensure accurate evaluations of follow-up pain and wound healing

In the intervention group:

1. Following the local anaesthetics administration for the Soft tissue trimmer(STT) gingivectomies, Soft tissue trimmer will be used with 400-rpm rotary systems and with no serum irrigation, per the manufacturer's recommendation.
2. Gingivoplasties will be performed with the same Soft tissue trimmer to easily provide a knife-edge appearance.
3. No periodontal packs will be applied to ensure accurate evaluations of follow-up pain and wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Anterior region (minimum of four teeth at each surgical site)
* Age range (18-45) years old
* Plaque-induced inflammatory gingival enlargement
* Altered passive eruption
* No clinical attachment loss
* Systemically healthy individuals

Exclusion Criteria:

* Gingival enlargement due to any systemic predisposing factors
* Pregnancy and/or lactation
* Allergy
* Conditions requiring antibiotic prophylaxis and anti-inflammatory medications.
* Acute or untreated periodontitis
* Systemic disease that could influence the outcome of the treatment (i.e. Diabetes)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Pain VAS | 7 days
  Visual Analogue Scale for Pain (numbers from 0 to 10 ('no pain' to 'worst pain imaginable') measured 1,3,5 and 7 days postoperatively.

SECONDARY OUTCOMES:
Epithelization | 14 days.
  Re-epithelization after removal of excess tissue will be assessed either partial or complete.This will be tested by toluidine blue (TB)
Tissue colour | 6 weeks.
  If it is either redder or whiter than the opposite side, or like opposite side tissue.
Bleeding | From 3-5 days
  If bleeding spontaneously or on palpation exists or not.
Surgical time | During surgical procedure itself.
  Time taken for both groups of surgery( control and intervention) will be measured from the administration of anaesthesia till removal of excess tissues.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine-CU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes